CLINICAL TRIAL: NCT03999684
Title: A Phase II Trial of All-trans Retinoic Acid (ATRA) in Advanced Adenoid Cystic Carcinoma
Brief Title: A Trial of All-trans Retinoic Acid (ATRA) in Advanced Adenoid Cystic Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: The V Foundation (Other); Adenoid Cystic Carcinoma Research Foundation (Other)
Responsible Party: Principal Investigator, Glenn J. Hanna, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-224
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Results first posted 2021-08-06 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Adenoid Cystic Carcinoma
Keywords: Adenoid Cystic Carcinoma
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tretinoin (Experimental): -Participants will receive Tretinoin orally divided over two daily doses for days 1 through 14 of a 28-day cycle
  Interventions: Drug: Tretinoin

INTERVENTIONS:
Drug: Tretinoin — ATRA control normal cell growth, cell differentiation (the normal process of making cell different from each other), and cell death during embryonic development and in certain tissues later in life. Retinoids effects on the cells are controlled by receptors on the nucleus of each cell (nuclear receptors)
  Other Names: Tretin-X; ATRA

SUMMARY:
This research is studying how safe and effective all-trans retinoic acid (ATRA), is to treat advanced adenoid cystic carcinoma (ACC).

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved all-trans retinoic acid (ATRA) for this specific disease but it has been approved for other uses.

The main purpose of this study is to see how effective all-trans retinoic acid (ATRA) is in treating tumor. Other reasons for conducting the study are:

* To determine for how long all-trans retinoic acid (ATRA) may reduce the size or slow down the growth of tumor
* To evaluate levels of circulating tumor DNA (ctDNA) released in the bloodstream as an indication of the disease activity
* To better understand mechanisms of tumor resistance to ATRA

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed adenoid cystic carcinoma with evidence of recurrent, metastatic or advanced, unresectable disease that is not amenable to curative surgery with or without radiotherapy.
* Participants must have at least one RECIST v1.1 measurable non-CNS based lesion, as defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) equal to or greater than 1 cm with CT scans or MR imaging.
* Participants must be willing to undergo fresh tissue core needle biopsy prior to study registration and repeat tumor biopsy while on study for correlatives. Willingness to provide blood samples for research throughout the study is also required.
* Prior systemic therapy: At least 2 weeks must have elapsed since the end of prior chemotherapy, biological agents (4 weeks for anti-cancer monoclonal antibody containing regimens) or any investigational drug product, with adequate recovery of treatment-related toxicity to NCI CTCAE Version 5.0 grade ≤ 1 (or tolerable grade 2) or back to baseline (except for alopecia or neuropathy). Any number of prior therapies for recurrent/metastatic ACC are permitted.
* Be ≥ 18 years of age on day of signing informed consent.
* Have a performance status of 0 or 1 on the ECOG Performance Scale (see Appendix A).
* Participants must have documentation of a new or progressive lesion on a radiologic imaging study performed within 12 months prior to study registration (progression of disease over any interval is allowed) and/or new or worsening disease-related symptoms within 12 months prior to study registration. This assessment is performed by the treating investigator. Evidence of progression by RECIST v1.1 criteria is not required.
* Participants must have normal organ and marrow function as defined below (within 14 days prior to study registration):

  * leukocytes ≥ 3,000/mcL
  * absolute neutrophil count ≥ 1,500/mcL
  * hemoglobin ≥ 9 g/dL without transfusion within 7 days of treatment
  * platelets ≥ 100,000/mcL
  * total bilirubin ≤ 2x upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤ 2.5x institutional ULN or ≤ 5x ULN for those with liver metastases
  * serum creatinine ≤ 1.5x ULN OR
  * creatinine clearance ≥ 60 mL/min/1.73 m2 for participants with creatinine levels above 1.5x ULN
  * coagulation profile INR ≤ 1.5x ULN unless the participant is receiving an anticoagulant
  * triglyceride level < 500 mg/dL or < 5.7 mmol/L
  * cholesterol level < 400 mg/dL or < 10.34 mmol/L
* Baseline tumor measurements must be documented from imaging within 28 days prior to study registration. Other non-laboratory tests must be performed within 28 days prior to study registration.
* Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 14 days of study registration. Female subjects of childbearing potential should have a negative urine or serum pregnancy test repeated within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female and male subjects of childbearing potential must agree to use an adequate method of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 4 months after completion of tretinoin administration. Contraception is required before starting the first dose of study medication through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject. There is a significant risk of fetal malformation if pregnancy occurs while on tretinoin at any dose level, even if for short exposure periods.
* Be willing and able to provide written informed consent for the trial.

Exclusion Criteria:

* Metastatic disease impinging on the spinal cord or threatening spinal cord compression. Patients that have had previous treatment of disease with impinging on the cord with either surgery or radiotherapy with clinical or radiographic evidence of response or stability are eligible.
* Participant has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment), and have no evidence of new or enlarging brain metastases. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability, because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Concurrent administration of other cancer specific therapy or investigational agents during the course of this study is not allowed.
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Subjects who are pregnant, or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment. Pregnant women are excluded from this study because tretinoin has the potential for teratogenic or abortifacient effects. Breastfeeding should be discontinued if the mother is treated on this protocol. Women who could potentially become pregnant while undergoing treatment on this protocol must be willing to use 2 methods of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J. Hanna, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tretinoin
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tretinoin
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 58 [40 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 17
  Other | 1
  Non-Hispanic | 18
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate
Description: CR 0, PR 0, SD 11, PD 5, UE 2
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. SD=stable disease, PD=progression of disease, UE=unevaluable
Time Frame: up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tretinoin
Number analyzed (Participants) | 18
Participants
  CR | 0
  PR | 0
  SD | 11
  PD | 5
  UE | 2

2. Secondary Outcome: Complete Response
Description: CR rate captured up to 8 months
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. SD=stable disease, PD=progression of disease, UE=unevaluable
Time Frame: up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tretinoin
Number analyzed (Participants) | 18
Participants | 0

3. Secondary Outcome: Partial Response
Description: PR rate captured up to 8 months
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. SD=stable disease, PD=progression of disease, UE=unevaluable
Time Frame: up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tretinoin
Number analyzed (Participants) | 18
Participants | 0

4. Secondary Outcome: Progression Free Survival
Description: Median PFS or progression free survival
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. SD=stable disease, PD=progression of disease (Progression was defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions), UE=unevaluable
Time Frame: up to 8 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tretinoin
Number analyzed (Participants) | 18
months | 3.2 [1.8 to 3.9]

5. Secondary Outcome: Duration Of Therapeutic Response
Description: Duration of CR+PR
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. SD=stable disease, PD=progression of disease, UE=unevaluable
Time Frame: up to 8 months
Measure: Median (Full Range); unit: months
Arm/Group | Tretinoin
Number analyzed (Participants) | 18
months | NA [NA to NA] — No participants showed any complete or partial response

6. Other Pre Specified Outcome: Number of Participants With no/Low, Medium MYB Expression in ACC Tumors
Description: correlative measure of ATRA inhibitory effect measured by IHC (units: % MYB inhibition by IHC quantitative measurement; MYB IHC was performed on stained tissue slides from baseline tumors and scored (%) by an expert pathologist as no/low, medium, and high MYB expressing).
Time Frame: up to 8 months
Population: only 14 patients had samples evaluable for MYB IHC assessment (of a total of 18)
Measure: Count of Participants; unit: Participants
Arm/Group | Tretinoin
Number analyzed (Participants) | 14
Participants
  Low MYB expression | 3
  Medium or high MYB expression | 11

ADVERSE EVENTS:
Time Frame: 8 months
Description: No difference
Arm/Group | Tretinoin
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 14/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tretinoin (N=18)
Dry Skin (Skin and subcutaneous tissue disorders) | 14
Headache (General disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-31): https://cdn.clinicaltrials.gov/large-docs/84/NCT03999684/Prot_002.pdf
  • Statistical Analysis Plan (2019-12-31): https://cdn.clinicaltrials.gov/large-docs/84/NCT03999684/SAP_004.pdf